CLINICAL TRIAL: NCT02055872
Title: A Single-centre, Randomized, Double-blinded, Placebo-controlled Pilot Study to Determine the Feasibility of a Full-scale Clinical Trial to Compare the Effect of Furosemide With or Without 25% Albumin in the Diuresis of Edema in Volume-overloaded ICU Patients in the Post-resuscitation Phase of Illness.
Brief Title: Furosemide and Albumin for Diuresis of Edema: A Pilot Randomized Controlled Trial
Acronym: FADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIF-13343
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-09

CONDITIONS: Edema; Hypoproteinemia
Keywords: Edema; Hypoproteinemia; Albumin; Diuresis; Critical illness
MeSH Terms: conditions — Edema; Hypoproteinemia; Critical Illness | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous albumin (Experimental): Administration of 25% albumin by intravenous infusion, twice daily for a total of 72 hours (6 treatments)
  Interventions: Drug: Intravenous albumin
- Normal saline (Placebo Comparator): Administration of 100 mL normal saline by intravenous infusion, twice daily, for 72 hours (6 treatments)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Intravenous albumin
  Arms: Intravenous albumin
Drug: Normal saline
  Arms: Normal saline

SUMMARY:
Critically ill patients usually require intravenous fluids to correct low blood pressure and improve blood flow to vital organs. However, once the patient's blood pressure has improved, these fluids can leak out into various organs, including the lung, kidneys, and skin. Excess fluid in these tissues, called edema, has been associated with longer ICU stays and higher mortality. Thus removing excess fluid is an important goal. The simplest way to treat edema is to use diuretics, such as furosemide, which increase urine output.

To further improve urine output, patients are sometimes given albumin, a protein which helps to suck fluid out from the tissues, and keep it in the blood vessel, where it can be filtered in the kidney and removed in the urine. Although albumin is often used for this purpose, there is little evidence to support it. A large randomized controlled trial is needed to determine if albumin plus furosemide is truly more effective than furosemide alone in critically ill patients with low levels of blood albumin. We will perform a pilot study to assess the feasibility of such a trial.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable for at least 24 hours (absence of persistent [>1 h] hypotension [systolic blood pressure <90 mmHg), not currently on vasopressors, less than 2 L crystalloid or colloid boluses, or 2 units red blood cells administered, maintenance fluids excluded
* Hypoproteinemia (serum albumin <30 mg/L or total protein < 60 mg/L)
* Clinical decision to diurese at least 3 L net fluid balance within the next 72 hours for any reason

Exclusion Criteria:

* known pregnancy
* patient or surrogate unable or unwilling to consent to blood product administration, including albumin
* history of adverse reactions or allergy to either albumin or furosemide
* acute kidney injury (RIFLE criteria "F" or greater) without any improvement in past 24 hours, or otherwise expected to necessitate dialysis within 48 hours in opinion of treating physician
* chronic kidney injury requiring dialysis
* clinically documented cirrhosis
* clinically documented nephrotic syndrome
* serum sodium greater than 150 milliequivalent/L or serum potassium less than 2.5 mEq/L that connote be treated prior to administration of study treatment
* inability to measure urine output and fluid balance
* Receipt of hyperoncotic albumin within preceding 24 hours
* previous enrollment in this trial, or any research studies which may interfere with this study
* estimated survival or ICU stay less than 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Oczkowski, MD, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Oczkowski SJ, Mazzetti I, Meade MO, Hamielec C. Furosemide and albumin for diuresis of edema (FADE): a study protocol for a randomized controlled trial. Trials. 2014 Jun 12;15:222. doi: 10.1186/1745-6215-15-222. PMID 24919684

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Albumin (n=24): Administration of 25% albumin by intravenous infusion, twice daily for a total of 72 hours (6 treatments)
  Intravenous albumin
- Normal Saline (n=21): Administration of 100 mL normal saline by intravenous infusion, twice daily, for 72 hours (6 treatments)
  Normal saline
Period: Overall Study
Arm/Group | Intravenous Albumin (n=24) | Normal Saline (n=21)
Started | 24 | 21
Completed | 24 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Albumin (n=24) | Normal Saline (n=21) | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.71 (17.2) | 64.7 (15.2) | 63.1 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days
Description: Ventilator-free days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intravenous Albumin (n=24) | Normal Saline (n=21)
Number analyzed (Participants) | 24 | 21
days | 4 [0 to 23.5] | 13 [0 to 21]

2. Secondary Outcome: Serum Albumin and Colloid Osmotic Pressure
Description: Changes in serum albumin and serum colloid osmotic pressure measurements from Day 1, Day 3, Day 5
Time Frame: Day 1, Day 3, Day 5
Reporting Status: Not Posted

3. Secondary Outcome: Mortality
Description: Total ICU mortality and mortality at 30 days.
Time Frame: 30 days
Reporting Status: Not Posted

4. Secondary Outcome: Fluid Balance and Body Weight
Description: Change in total fluid balance and body weight from baseline at 3 days and 5 days
Time Frame: Day 1, Day 3, Day 5
Reporting Status: Not Posted

5. Secondary Outcome: Oxygenation
Description: Changes in oxygenation (FiO2, P/F ratio, oxygenation index) from baseline at day 3 and day 5
Time Frame: Day 1, Day 3, Day 5
Reporting Status: Not Posted

6. Secondary Outcome: Treatment Interruptions
Description: Number of episodes of interrupting treatment with furosemide (eg. hypotensive episodes, renal failure, contraction alkalosis, etc.)
Time Frame: Day 1, Day 2, Day 3
Reporting Status: Not Posted

7. Secondary Outcome: Duration of Mechanical Ventilation
Description: Total duration of mechanical ventilation
Time Frame: 30 days
Reporting Status: Not Posted

8. Secondary Outcome: Length of ICU Stay
Time Frame: Study end
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Adherence to Protocol
Description: The administration of at least the first dose of study treatment (albumin or placebo) within two hours of the first administration of furosemide
Time Frame: Day 1
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Completion of Study Treatment
Description: Patients receiving full 72 hours (6 doses) of study treatment
Time Frame: Day 3
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Absence of Co-intervention
Description: Absence of hyperoncotic albumin administration to patients randomized to the control arm
Time Frame: Day 3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Randomization Rate
Description: 1. Randomization rate of patients eligible by screening criteria
  2. Randomization rate of patients eligible by clinical site
Time Frame: Study duration
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intravenous Albumin (n=24) | Normal Saline (n=21)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 2/24 | 4/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Albumin (n=24) (N=24) | Normal Saline (n=21) (N=21)
Hypotension (Cardiac disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes